CLINICAL TRIAL: NCT03283917
Title: A Safety Study of Daratumumab, Ixazomib, and Dexamethasone in AL Amyloidosis
Brief Title: Daratumumab, Ixazomib, and Dexamethasone in AL Amyloidosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0243; NCI-2018-01044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0243 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Newly Diagnosed Primary Amyloidosis; Recurrent Primary Amyloidosis; Refractory Primary Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; MLN2238

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab, ixazomib, dexamethasone) (Experimental): Participants receive daratumumab IV over 3.5-6.5 hours on days 1, 8, 15, and 22 of courses 1-2, on days 1 and 15 of courses 3-6, and on day 1 of courses 7-12. Participants also receive ixazomib PO on days 1, 8, and 15, and dexamethasone IV over 15 minutes or PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unaccepted toxicity.
  Interventions: Biological: Daratumumab; Drug: Dexamethasone; Drug: Ixazomib

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib — Given PO
  Other Names: MLN-2238; MLN2238

SUMMARY:
This phase I trial studies the side effects and best dose of daratumumab, ixazomib, and dexamethasone in treating participants with amyloid light chain amyloidosis. Monoclonal antibodies, such as daratumumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as ixazomib and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving daratumumab, ixazomib, and dexamethasone may be effective in treating participants with light chain amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm the safety and tolerability of daratumumab, ixazomib, and dexamethasone (DId) in patients with amyloid light chain (AL) amyloidosis.

II. To determine the recommended phase 2 dose (RP2D) of daratumumab, ixazomib, and dexamethasone in subjects with AL amyloidosis.

SECONDARY OBJECTIVES:

I. To determine the hematologic response rate of daratumumab, ixazomib, and dexamethasone in patients with AL amyloidosis.

II. To determine cardiac and renal organ response rate of daratumumab, ixazomib, and dexamethasone in patients with AL amyloidosis.

III. To determine time to next therapy. IV. To determine the time to response. V. To determine the duration of response. VI. To determine progression free survival (PFS). VII. To determine overall survival (OS).

OUTLINE: This is a dose-escalation study of dexamethasone.

Participants receive daratumumab intravenously (IV) over 3.5-6.5 hours on days 1, 8, 15, and 22 of courses 1-2, on days 1 and 15 of courses 3-6, and on day 1 of courses 7-12. Participants also receive ixazomib orally (PO) on days 1, 8, and 15, and dexamethasone IV over 15 minutes or PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, participants are followed up at 30 days and then every 90 days for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary systemic AL amyloidosis of tissue as determined by: a. Congo red staining of tissue showing apple green birefringence AND b. Clonal plasma cell disorder as determined by: i. Immunohistochemistry, in situ hybridization (ISH) or flow cytometry demonstrating kappa or lambda light chain restriction on bone marrow biopsy AND/OR ii. Monoclonal protein on serum or urine electrophoresis/immunofixation OR abnormal free light chain ratio
* Newly diagnosed OR relapsed and/or refractory AL amyloidosis. Newly diagnosed patients must be treatment naive without previous plasma cell-directed therapy with the exception of a maximum of 160 mg dexamethasone or equivalent prior to dosing on protocol. Relapsed and/or refractory is defined as follows: a. Clonal relapse after at least one previous line of therapy or high-dose chemotherapy and autologous stem cell transplantation OR b. Refractory disease to prior therapy defined as less than a hematologic very good partial response (VGPR). If previous therapy was autologous stem cell transplant (SCT), must be >= 3 months after SCT
* Measurable disease defined by: a. Monoclonal protein in the serum or urine by immunofixation OR plasmacytosis of bone marrow with monoclonal staining for kappa or lambda light-chain isotype b. dFLC >= 50 mg/L (dFLC=difference in involved and uninvolved serum free light-chain levels)
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 75,000/mm^3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 10 mL/min

Exclusion Criteria:

* Non-AL amyloidosis
* Clinically overt myeloma a.) Lytic bone lesions or biopsy proven plasmacytoma b.) Hypercalcemia (corrected for albumin) > 11 mg/dL unexplained by other causes
* Clinically significant cardiac disease defined by any of the following criteria: a.) New York Heart Association (NYHA) class IV heart failure b.) N-terminal prohormone of brain natriuretic peptide (NT-ProBNP) > 8500 ng/L c.) Symptomatic orthostatic hypotension with supine systolic blood pressure < 90 mm Hg d.) Unstable cardiac arrhythmia e.) Unstable angina f.) Myocardial infarction within the past 6 months
* Severe obstructive airway disease defined by forced expiratory volume at one second (FEV1) < 50%
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (ie, =< grade 1 toxicity) from the reversible effects of prior chemotherapy
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Infection requiring systemic intravenous antibiotic therapy or other serious infection within 14 days before study enrollment
* Systemic treatment, within 14 days before the first dose of and dexamethasone (DId), with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Patients that have previously been treated with daratumumab or ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2027-05-18 (Estimated); Study Completion 2027-05-18 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rate | Up to 28 days
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.
Recommended phase 2 dose of daratumumab, ixazomib, and dexamethasone | Up to 24 months

SECONDARY OUTCOMES:
Overall hematologic response rate | Up to 24 months
Time to response | Up to 24 months
Duration of response | Up to 24 months
Time to next therapy | Up to 24 months
Progression free survival | Up to 24 months
Overall survival | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org